CLINICAL TRIAL: NCT01636700
Title: Comparative Study of Analgesic Effect and Serum IL-6 With Tramadol Infiltration or Intravenous After Tonsillectomy
Brief Title: Tramadol Infiltration for Tonsillectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rioko Kimiko Sakata, Pain Clinic Director, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP2011
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2014-02

CONDITIONS: Postoperative Pain
Keywords: Tramadol infiltration; Analgesic effect; Serum IL-6
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol; Analgesics, Opioid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tramadol infiltration (Active Comparator): infiltration of tramadol 2mg/kg
  Interventions: Drug: Tramadol 2mg/kg
- Saline solution (Placebo Comparator): Infiltration of saline
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Tramadol 2mg/kg — 2mg/kg
  Other Names: Opioid
  Arms: tramadol infiltration
Drug: Saline solution — saline solution- 1 dose
  Other Names: Placebo
  Arms: Saline solution

SUMMARY:
The purpose of this study is to evaluate the analgesic effect and IL-6 after tramadol infiltration or intravenous for tonsillectomy.

DETAILED DESCRIPTION:
The study will be prospective, double-blind, randomized study of 40 children aged ≥ 4 and ≤ 12 years undergoing tonsillectomy under general anesthesia.

Patients will be allocated into two groups. Group 1 patients will receive tramadol 2 mg / kg intravenously and saline 0.9% infiltration in tonsils; group 2, will receive tramadol 2 mg / kg infiltration and intravenous saline.

There will be evaluated: postoperative pain intensity by facial scale, supplementary analgesics and interleukin-6. For statistical analysis of the results will be used parametric and nonparametric tests, taking into account the nature of the variables. The level of statistical significance will be set at < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* children aged ≥ 4 and ≤ 12 years undergoing tonsillectomy

Exclusion Criteria:

* coagulopathy,
* cancer,
* hepatic or renal alteration

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Analgesic effect | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, Study Director — Universidade Federal de São Paulo
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil